CLINICAL TRIAL: NCT06689449
Title: Comparison Effects of Erector Spinae Plan Block(ESP), Paravertebral Block(PVB) and Mid-point Transverse Process to Pleura Block(MTP) on Perioperative Pain Measured With Analgesia Nociceptive Index Monitor on Video-assisted Thoracoscopic Surgey(VATS)
Brief Title: Comparison Effects of Three Regional Anesthetic Technique on Pain During Video-assisted Thorascopic Surgery(VATS)
Status: Active, not recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Recep Aksu, clinical Professor.Recep AKSU, TC Erciyes University
Other Study IDs: 2024/165
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Video Assisted Thoracic Surgery (VATS)
Keywords: video assisted thoracic surgery; erector spinae plan block; paravertebral block; mid-point transverse process to pleura block; analgesia nosiseption index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- erector spinae plan block group: The patient will be monitored with routine monitoring and ANI under operating room conditions. VAS values and vital signs before and after peripheral nerve block will be recorded. Patients will be placed in the lateral position and an erector spinae plane block will be applied under USG guidance by an experienced anesthesiologist. Surgery will be allowed 30 minutes after the block is performed.
- paravertebral block group: The patient will be monitored with routine monitoring and ANI under operating room conditions. VAS values and vital signs before and after peripheral nerve block will be recorded. Patients will be placed in the lateral position and a paravertebral block will be applied under USG guidance by an experienced anesthesiologist. Surgery will be allowed 30 minutes after the block is performed.
- mid-point transverse process to pleura block group: The patient will be monitored with routine monitoring and ANI under operating room conditions. VAS values and vital signsbefore and after peripheral nerve block will be recorded. Patients will be placed in the lateral position and a mid-point transverse process to pleura block will be applied under USG guidance by an experienced anesthesiologist. Surgery will be allowed 30 minutes after the block is performed.

SUMMARY:
In this study, our iş to compare effect of erector spinae plan block(ESP), paravertebral block(PVB) and mid-point transverse process to pleura block(MTP) on perioperative pain measured with analgesia nociceptive index monitor on video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive thoracic surgery procedure performed with the help of a retractor-free camera through small skin incisions used to diagnose and treat chest diseases. Many of the major procedures traditionally performed with open thoracoscopic surgery can be performed using smaller sections with video assistance.

Thanks to the advances in minimally invasive techniques, the non-intubated thoracoscopic approach has been adapted even for use with major lung resections.

An adequate analgesia obtained from regional anaesthesia techniques allows VATS to be performed in sedated patients and the potential adverse effects related to general anaesthesia and selective ventilation can be avoided. The non-intubated procedures try to minimize the adverse effects of tracheal intubation and general anaesthesia, such as intubation-related airway trauma, ventilation-induced lung injury, residual neuromuscular blockade, and postoperative nausea and vomiting.

Local anaesthetic techniques essential for nonentubeted video assisted thoracic surgery include thoracic epidural anaesthesia, cervical epidural anaesthesia, paravertebral block, intercostal nerve block, injection of local anaesthetic at the site of trocar incision local vagus blockade, erector spinae plane block, serratus anterior plane block and pectoralis nerve block.

Thoracic epidural analgesia, once considered the gold standard for thoracotomy; due to the risks of complications related to dural puncture, epidural hematoma, neuropathy and hypotension, it is no longer the first choice for VATS and has been replaced by peripheral blocks.

ANI is a monitor that can be measured continuously and non-invasively. It measures parasympathetic tone - based on electrocardiography - by analyzing minimal changes in heart rate that occur under anesthesia, in the early stages of awakening, and in each respiratory cycle of awake patients. At the end of the measurement, a value between 0-100 is obtained.

Parasympathetic modulation (stress level, e.g., pain) is obtained with a minimum value of 0 and a maximum of 100. ANI values measured in the early period of recovery correlate with pain scores. When compared with hemodynamic parameters, it has been reported that the ANI response is more sensitive to nociceptive stimuli occurring in the intraoperative period.

In the high-risk patient group who will undergoing video-assisted thoracoscopic surgery (VATS) in the Faculty of Medicine of Erciyes University, the pain sensation in patients will be evaluated using ANI in the perioperative period, after the peripheral nerve blocks have been applied to different anatomical areas that are routinely used.

The aim of this study is to objectively reveal the perioperative pain after peripheral block applications in the patient group with serious additional morbidities by using the ANI device. It is expected that this study will enable more effective analgesia control in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18 under the 80 Who will undergo video assisted thoracic surgery -ASA group 2-3-4.
* Patients without opioid addiction.
* Patients without allergies.
* Patients without psychiatric disorder.
* Patients without arrhymia and beta-blocker use.
* Patients without contraindications for peripheral blocks.

Exclusion Criteria:

* Patients under age of 18
* Patients undergo surgery under general anesthesia
* Patients undergo emergency surgery
* Patients allergic to local anesthesia
* Patients wit bleeding diathesis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ASA group 2-3-4 patients older than 18 years of age who will under go video assisted thoracic surgery
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Effective analgesia control in patients with Analgesia Nociception Index(ANI) | intraoperative
  With Analgesia Nociception Index (ANI), it is advantageous to evaluate the objective findings measuring parasympathetic system activity. ANI is a monitor that can be measured continuously and non-invasively. It measures parasympathetic tone - based on electrocardiography - by analyzing minimal changes in heart rate that occur under anesthesia, in the early stages of awakening, and in each respiratory cycle of awake patients. A value between 0-100 is obtained, Values between 50 and 70 indicate good analgesia control. According to studies on ANI, the patient feels pain below 50. If it is above 70, it means that more analgesia is provided. It is thought that pain control will be more effective with these objective data.

SECONDARY OUTCOMES:
Visual analog scale | ıntraoperative and postoperative 24 hour
  A Visual Analogue Scale (VAS) is one of the pain rating scales. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest the VAS score for grading of pain consists of a 10 centimetres (cm) line with 10 mm (0.01 cm) to each point of the scale and two end-points representing no pain and worst possible pain, where 0 = no pain, 1-3 = mild, 4-6 = moderate and 7-10 = severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Recep aksu, Kayseri, Kayseri̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No